CLINICAL TRIAL: NCT02493920
Title: Evaluation of Pulmonary Mechanics in Preterm Infant Treated With Sustained Lung Inflation at Birth
Brief Title: Sustained Lung Inflation and Pulmonary Mechanics in Preterm Infant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems, unreliability of the measured parameters
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Mariarosa Colnaghi, Medical doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MECCANICA SLI
Record Dates: First submitted 2015-06-23; First posted 2015-07-10 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Preterm Birth; Respiratory Distress Syndrome; Lung Diseases
Keywords: Respiratory Distress Syndrome, Newborn; Delivery Room; Resuscitation; Premature birth; Infant, Newborn; Respiration Artificial
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Lung Diseases; Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLI group (Experimental): In this group the preterm infants will receive sustained lung inflation (SLI) with mask in the delivery room; the parameters of respiratory mechanics will be monitored for 5 minutes by means of the forced oscillation technique.
  Interventions: Other: Sustained lung inflation; Device: mask using a T-piece system (Fabian,Acutronic Medical Systems AG, Switzerland).
- Control (No Intervention): Preterm infants will be assisted in the delivery room with a continuous positive airway pressure (CPAP) of 5 cmH2O with mask and the parameters of respiratory mechanics will be monitored for 5 minutes by means of the forced oscillation technique.

INTERVENTIONS:
Other: Sustained lung inflation — Sustained lung inflation (SLI) will be performed with mask using a T-piece system (Fabian,Acutronic Medical Systems AG, Switzerland).Peak inflation pressure (PIP) of 25 cm H2O will be delivered for 15 seconds and then reduced to a PEEP of 5 cm H2O. A second SLI manoeuvre will be repeated in case of persistent hearth failure (HR <100 bpm).
  Other Names: lung recruitment
  Arms: SLI group
Device: mask using a T-piece system (Fabian,Acutronic Medical Systems AG, Switzerland).
  Arms: SLI group

SUMMARY:
Lung protection should start in the delivery room where, from the first breaths, the preterm infant can be helped to clear the lung fluid and to recruit alveolar spaces and establish the functional residual capacity (FRC). Sustained lung inflation (SLI) applied at birth in the delivery room has been demonstrated to lead to clearance of lung fluid and achievement of a precocious functional residual capacity (FRC) both in animal and human studies. SLI associated to an adequate positive end expiratory pressure (PEEP) may help the efficacy of the respiratory effort in lung of preterm infants at risk for respiratory distress syndrome (RDS) and reduce need of mechanical ventilation (MV).

Further studies are required to evaluate the clinical utility of this maneuver. The ability to monitor what happens to the lungs while applying different recruitment maneuvers in preterm infants would allow the definition of a procedure that allows optimal assistance to improve the FRC. One promising approach is provided by the forced oscillation technique (FOT). During forced oscillations, a small amplitude sinusoidal pressure stimulus is applied to the airway opening and the mechanical response of the respiratory system is studied by means of the total respiratory input impedance (Zin). Zin is a complex number that can be expressed as real part, called resistance (Rrs), and imaginary part, called reactance (Xrs). Particularly, it has been recently shown that Xrs measured at 5 Hz is very sensible to changes in the mechanics of lung periphery and provides accurate information about lung volume recruitment and derecruitment. The main purpose of this work is to apply FOT to the assessment of lung function in newborns submitted to SLI at birth. The investigators hypothesized that the application in the delivery room of the SLI in the preterm infant is effective in achieving a greater FRC and therefore a greater value of Xrs compared to a control group not treated with the SLI.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) at least 25 weeks but less than 36 completed weeks by best obstetrical estimate

Exclusion Criteria:

* Refusal of antenatal informed consent
* Known major anomalies, pulmonary hypoplasia
* Severe perinatal suffering

Ages: 25 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Estimated); Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in Reactance (Xrs) values measured by the forced oscillation technique (FOT) | Baseline and at 5 minutes of life (that is, before and at the end of the SLI)

SECONDARY OUTCOMES:
Need for intubation within the first 72 hours of life | 72 hours of life
Duration of respiratory support (ventilation, CPAP, supplemental oxygen) | During hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Death in hospital | During hospitalization - up to 40 weeks Post Menstrual Age (PMA)
Number of surfactant doses | During hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Retinopathy of prematurity (ROP) stage 3 or greater requiring treatment | 40 weeks Post Menstrual Age (PMA)
Incidence of Patent Ductus Arteriosus (PDA) requiring treatment | During hospitalization - up to 36 weeks Post Menstrual Age (PMA)
Incidence of Bronchopulmonary dysplasia | 36 weeks Post Menstrual Age (PMA)
  Defined according to the criteria of Jobe and Bancalari (Jobe A, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med 2001;163:1723-9)
Incidence of Intracranial Hemorrhages (ICH) | During hospitalization- up to 40 weeks Post Menstrual Age (PMA)
  We used the ICH classification of Papile et al
Length of hospital stay | Average discharge between 36 - 40 weeks PMA

CONTACTS AND LOCATIONS:
Overall Officials: Mariarosa Colnaghi, MD, Principal Investigator — NICU, IRCCS Cà Granda, Ospedale Maggiore Policlinico, Milan